CLINICAL TRIAL: NCT03862859
Title: The Danish Warfarin-Dialysis Study: Safety and Efficacy of Warfarin in Patients With Atrial Fibrillation on Dialysis - A Nationwide Parallel-group Open Randomized Clinical Trial
Brief Title: The Danish Warfarin-Dialysis Study - Safety and Efficacy of Warfarin in Patients With Atrial Fibrillation on Dialysis
Acronym: DANWARD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nicholas Carlson (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Sponsor-Investigator, Nicholas Carlson, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DANWARD 1.26; 2018-000484-86 (EudraCT Number)
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation and Flutter; Stroke; Major Bleed; End-stage Renal Disease
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Kidney Failure, Chronic | interventions — Warfarin; Vitamin B 6

STUDY DESIGN:
Intervention Model Description: A multicentre, randomized, open label, parallel group study.
Masking Description: None (Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Warfarin (Active Comparator): Warfarin with dosing targeting an international normalized ratio of 2-3.
  Interventions: Drug: Warfarin
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Drug: Warfarin — Dose adjusted Warfarin targeting an international normalized ratio of 2-3.
  Other Names: Coumadin; Marevan; Jantoven
  Arms: Treatment with Warfarin

SUMMARY:
The study aims to evaluate the appropriateness of initiating oral anticoagulation for stroke risk reduction in dialysis populations with atrial fibrillation. Specifically, the study will assess the overall safety, tolerability, and efficacy of initiating treatment with Warfarin in patients with end-stage renal disease on dialysis and atrial fibrillation.

DETAILED DESCRIPTION:
Data pertaining to the tolerability, safety, and benefit of initiating anticoagulation for stroke risk reduction in patients with end-stage renal disease and atrial fibrillation remains conflicting and insufficient. Patients on dialysis continue to be routinely excluded from randomized controlled trials, and evidence from observational studies is plausibly biased. The main objective of the following parallel-group open randomized clinical trial presents a nationwide study aimed at investigating the benefit, tolerability, and safety of initiating warfarin versus no treatment in patients with atrial fibrillation on dialysis. The anticipated results from this project will provide conclusive evidence as to the appropriateness of initiating oral anticoagulation for stroke risk reduction in dialysis populations with atrial fibrillation with direct effects on clinical management and international guidelines pertaining to these patients.

The study is planned as a multicentre, randomized, open label, parallel group trial with planned inclusion of a total of 718 patients (359 patients per arm). Dialysis-treated patients with end-stage renal disease with paroxysmal, persistent, or permanent atrial fibrillation will be enrolled and randomized to either treatment with warfarin or no treatment. Randomization with be attained using a 1:1 allocation as per a computer-generated randomization schedule stratified by gender, age by decade, and center using permuted blocks of random sizes. Study participants will be allocated to treatment in accordance with the randomization for the full duration of the trial i.e. at a minimum one year following randomization, and followed with regular monitoring for the the primary efficacy outcome of ischemic stroke or death due to ischemic or unspecified stroke and the primary safety outcome of major bleeding defined in accordance with the International Society on Thrombosis and Hemostasis definition.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years on chronic dialysis due to end-stage renal disease
* Non-valvular paroxysmal, persistent, or permanent atrial fibrillation OR non-treated (for >2 months) prevalent paroxysmal, persistent or permanent atrial fibrillation as documented by an electrocardiogram or an episode of ≥30 seconds on Holter monitor, or episodes ≥ 6 minutes on event recorders or any other recording device.
* Competence to understand the study rationale, including potential risks and benefits associated with treatment, necessary for written informed consent.

Exclusion Criteria:

* CHA2DS2-VASc Score ≤1
* Other indications for oral anticoagulation treatment (pulmonary embolism < 6 months, deep vein thrombosis <3 months, mechanical heart valve prosthesis) irrespective of whether treatment is implemented
* Ongoing dual antiplatelet treatment
* Malignancy (with exception of non-melanoma skin cancer) with recent < 1 year, ongoing, or planned curative, or palliative chemo- , radiation-, and/or scheduled surgical therapy
* Endoscopy with gastrointestinal ulcer <1 month
* Esophageal varices
* Autoimmune og genetic coagulation disorders
* Congenital alactasia, Lapp Lactase deficiency or glucose-galactose malabsorption
* Pending spinal tap
* Cerebrovascular malformations
* Arterial aneurysms
* Ulcers or wounds (Wagner grad >1)
* Bacterial endocarditis < 3 months
* Active bleeding contraindicating anticoagulation
* Any non-elective and/or non-ambulant surgery <7 days
* Cerebral hemorrhage <4 weeks
* Thrombocytopenia (platelet count <100 × 109/L) <30 days.
* Severe liver insufficiency (spontaneous international normalized ratio >1.5) <30 days.
* Known intolerance to warfarin
* Use of hypericum perforatum / St. John's Wort
* Uncontrolled hypertension (repeat blood pressure >180/110 mmhg) < 30 days
* Uncontrolled hyperthyroidism (thyroid-stimulating hormone <0.1μIU/mL) <30 days
* Pregnancy or lactation
* Participation in other ongoing intervention trials adjudged to influence study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome - Number of participants with transient ischemic attack, fatal and non-fatal ischaemic or unspecific stroke | From randomization to end of observation - up to 4 years
  Any transient ischemic attack, fatal and non-fatal ischaemic or unspecific stroke or death attributable to either ischemic or undefined stroke
Primary safety outcome - Number of participants with fatal or non-fatal major bleeding | From randomization to end of observation - up to 4 years
  Any major bleeding as defined in accordance with the International Society on Thrombosis and Hemostasis definition pertaining to major bleeding in non-surgical patients

SECONDARY OUTCOMES:
Number of participants with ischemic or unspecified stroke | From time of randomization to end of observation - up to 4 years
  Any non-fatal or fatal ischemic stroke or unspecified stroke event
Number of participants with ischemic stroke | From time of randomization to end of observation - up to 4 years
  Any non-fatal or fatal ischemic stroke event
Number of participants with hemorrhagic stroke | From time of randomization to end of observation - up to 4 years
  Any non-fatal or fatal hemorrhagic stroke event
Number of participants with ischemic or hemorrhagic stroke | From time of randomization to end of observation - up to 4 years
  Any non-fatal or fatal ischemic or hemorrhagic stroke event
Number of deaths | From time of randomization to end of observation - up to 4 years
  All-cause mortality
The combination of any non-fatal stroke and all-cause mortality | From time of randomization to end of observation - up to 4 years
  Number of participants with either non-fatal ischemic or hemorrhagic stroke of death due to any cause
The combination of any non-fatal stroke, any non-fatal major bleeding, and all-cause mortality | From time of randomization to end of observation - up to 4 years
  Number of participants with either non-fatal ischemic or hemorrhagic stroke, any non-fatal major bleeding as defined in accordance with the International Society on Thrombosis and Hemostasis definition pertaining to major bleeding in non-surgical patients, or death due to any cause

OTHER OUTCOMES:
Discontinuation of the allocated randomized therapy | From time of randomization to end of observation - up to 4 years
  Number of participants discontinuing the allocated randomized therapy irrespective of cause
Number of participants with peripheral artery disease | From time of randomization to end of observation - up to 4 years
  Any diagnosis of previously unverified peripheral artery disease
Number of participants with fatal or non-fatal acute myocardial infarction | From randomization to end of observation - up to 4 years
  Any non-fatal or fatal acute myocardial infarction event
Number of participants with calciphylaxis | From time of randomization to end of observation - up to 4 years
  Development of calciphylaxis as defined by clinical diagnosis
Number of participants hospitalized due to left-sided heart failure | From time of randomization to end of observation - up to 4 years
  Any hospitalization due to left-sided heart failure as defined by de novo LVEF <30% with echocardiographic verification
Percentage of participants with arteriovenous fistula thrombosis | From randomization to end of observation - up to 4 years
  Arteriovenous fistula thrombosis in participants dialyzed via an arteriovenous fistula
Number of participants with osteoporotic fractures | From randomization to end of observation - up to 4 years
  Osteoporotic fractures as defined by low energy fractures of the proximal femur, distal radius, humerus, pelvis, and vertebrae

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Carlson, MD PhD, Principal Investigator — Department of Nephrology, Copenhagen University Hospital Rigshospitalet; Gunnar H Gislason, Prof MD PhD, Study Chair — Danish Heart Foundation; Anne-Lise Kamper, MD DMSc, Study Chair — Department of Nephrology, Copenhagen University Hospital Rigshospitalet; Christian Torp-Pedersen, Prof MD DMSc, Study Chair — Department of Cardiology, North Zealand Hospital; Jonas B Olesen, MD PhD, Study Chair — Department of Cardiology, Copenhagen University Hospital Gentofte; Casper Bang, MD PhD, Study Chair — Department of Cardiology, Frederiksberg and Bispebjerg Hospital; Thomas A Gerds, Prof, Study Chair — Danish Heart Foundation; Ditte Hansen, MD PhD, Study Chair — Department of Nephrology, Copenhagen University Hospital Herlev; Morten Schou, Prof MD PhD, Study Chair — Department of Cardiology, Copenhagen University Hospital Herlev; Mads Hornum, Prof MD PhD, Study Chair — Department of Nephrology, Copenhagen University Hospital Rigshospitalet; Erik Grove, MD PhD, Study Chair — Department of Cardiology, Aarhus University Hospital; Jens D Jensen, MD PhD, Study Chair — Department of Nephrology, Aarhus University Hospital; Ellen Linnea F Ballegaard, MD, Study Chair — Department of Nephrology, Copenhagen University Hospital Rigshospitalet
Locations (13):
- Denmark (13):
  - Aalborg University Hosptial, Aalborg
  - Aarhus University Hospital, Aarhus
  - Department of Nephrology, Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Esbjerg and Grindsted Hospital, Esbjerg
  - Department of Nephrology, Herlev Hospital, Herlev
  - Department of nephrology, Nordsjaellands Hospital, Hillerød
  - Holbaek Hospital, Holbæk
  - Holstebro Hospital, Holstebro
  - Lillebælt Hospital, Kolding
  - Zealand University Hospital, Roskilde
  - Bornholms Hospital, Rønne
  - Hospital Sønderjylland, Sønderborg
  - Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcomes measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Data access requests will be reviewed, requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Ballegaard ELF, Lindhard K, Lindhardt M, Peters CD, Thomsen Nielsen F, Tietze IN, Borg R, Boesby L, Bertelsen MC, Brosen JMB, Cibulskyte-Ninkovic D, Rantanen JM, Mose FH, Kampmann JD, Nielsen AS, Breinholt JK, Kofod DH, Bressendorff I, Clausen PV, Lange T, Kober L, Kamper AL, Bang CNF, Torp-Pedersen C, Hansen D, Grove EL, Gislason G, Dam Jensen J, Olesen JB, Hornum M, Rix M, Schou M, Carlson N. Protocol for a randomised controlled trial comparing warfarin with no oral anticoagulation in patients with atrial fibrillation on chronic dialysis: the Danish Warfarin-Dialysis (DANWARD) trial. BMJ Open. 2024 Feb 26;14(2):e081961. doi: 10.1136/bmjopen-2023-081961. PMID 38413147